CLINICAL TRIAL: NCT05699278
Title: An Observational Study Evaluating The Experiences of Gastric Cancer Patients In Clinical Trials
Brief Title: Investigating the Experiences of Individuals With Gastric Cancer Participating in Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 87554209
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Gastric Cancer Stage
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is observational, meaning that it does not include any interventions or new treatments. As a result, there may not be an immediate benefit for the patient with gastric cancer.

However, the data collected from this trial can contribute to a better understanding of the factors that affect withdrawal and enrolment rates in gastric cancer clinical trials, and may ultimately lead to improved patient outcomes in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a minimum of 18 years or older
* Patient has been diagnosed with gastric cancer
* Patient has been self-identified as planning to enroll in an observational clinical study

Exclusion Criteria:

* Patient is breastfeeding or pregnant
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients who are actively considering participating in an observational clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a gastric cancer clinical trial | 3 months
Rate of patients who remain in a gastric cancer clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sexton RE, Al Hallak MN, Diab M, Azmi AS. Gastric cancer: a comprehensive review of current and future treatment strategies. Cancer Metastasis Rev. 2020 Dec;39(4):1179-1203. doi: 10.1007/s10555-020-09925-3. Epub 2020 Sep 7. PMID 32894370
- [Background] Mihaljevic AL, Friess H, Schuhmacher C. Clinical trials in gastric cancer and the future. J Surg Oncol. 2013 Mar;107(3):289-97. doi: 10.1002/jso.23120. Epub 2012 Apr 18. PMID 22514058
- [Background] Petryszyn P, Chapelle N, Matysiak-Budnik T. Gastric Cancer: Where Are We Heading? Dig Dis. 2020;38(4):280-285. doi: 10.1159/000506509. Epub 2020 Feb 17. PMID 32062657

DOCUMENTS (1):
  • Informed Consent Form (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT05699278/ICF_000.pdf